CLINICAL TRIAL: NCT03758131
Title: Peer-enhanced Motivational Interviewing in Federally-Qualified Health Clinics for Substance-using Emerging Adults
Brief Title: Peer MI in FQHCs for Substance-using Emerging Adults
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Smith17393FQHC
Record Dates: First submitted 2018-11-06; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Substance Use Disorders
Keywords: Motivational Interviewing
MeSH Terms: conditions — Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peer-enhanced Motivational Interviewing (Experimental): In the Peer-Enhanced Motivational Interviewing (PMI) condition, target clients and peers will receive separate one-hour sessions of Motivational Interviewing (MI), an empirically-supported treatment that helps individuals work through ambivalence about making changes in substance use. Mi is thought to work because it is a non-confrontational intervention where a therapist empathetically reviews substance use behaviors, listens empathetically, and reinforces any client statements indicating a desire to change. With the "peer" of each PMI dyad, the therapist presents peer with data about the extent of the target client's substance use, builds the peer's motivation to help their friend, and teaches the peer communication skills they can use to influence the target client's substance use.
  Interventions: Behavioral: Peer-enhanced Motivational Interviewing
- Motivational Interviewing (Active Comparator): In the Motivational Interviewing (MI) condition, target clients only will receive one-hour sessions of Motivational Interviewing (MI), an empirically-supported treatment that helps individuals work through ambivalence about making changes in substance use.
  Interventions: Behavioral: Motivational Interviewing
- Waitlist Control (Placebo Comparator): Those dyads randomized to the Waitlist Control (WC) condition willl be offered teh PMI intervention at month 2 post-intervention for the PMI arm.
  Interventions: Behavioral: Peer-enhanced Motivational Interviewing; Other: Waitlist Control

INTERVENTIONS:
Behavioral: Peer-enhanced Motivational Interviewing — In the Peer-Enhanced Motivational Interviewing (PMI) condition, target clients and peers will receive separate one-hour sessions of Motivational Interviewing (MI), an empirically-supported treatment that helps individuals work through ambivalence about making changes in substance use. MI is thought to work because it is a non-confrontational intervention where a therapist empathetically reviews substance use behaviors, listens empathetically, and reinforces any client statements indicating a desire to change. With the "peer" of each PMI dyad, the therapist presents peer with data about the extent of the target client's substance use, builds the peer's motivation to help their friend, and teaches the peer communication skills they can use to influence the target client's substance use.
  Other Names: PMI
  Arms: Peer-enhanced Motivational Interviewing; Waitlist Control
Behavioral: Motivational Interviewing — In the Motivational Interviewing (PMI) condition, target clients only will receive one-hour sessions of Motivational Interviewing (MI), an empirically-supported treatment that helps individuals work through ambivalence about making changes in substance use. MI is thought to work because it is a non-confrontational intervention where a therapist empathetically reviews substance use behaviors, listens empathetically, and reinforces any client statements indicating a desire to change.
  Other Names: MI
  Arms: Motivational Interviewing
Other: Waitlist Control — Dyads randomized to this intervention will have no contact with study personnel until 2 months after the PMI group has completed the PMI intervention. Then those in the Waitlist Control condition will receive the full PMI protocol.
  Other Names: WC
  Arms: Waitlist Control

SUMMARY:
The main purpose of this study is to test whether a Peer-Enhanced Motivational Interviewing (PMI) intervention, which has been successful with college students, results in superior alcohol and marijuana use outcomes for emerging adults (EA), ages 18-29, who are clients of Federally-qualified Health Centers, and their peers. In the first phase of the study, seventy-five peer dyads (total n = 150, ntarget client = 75, npeer = 75) will be randomized to receive either Peer-Enhanced Motivational Interviewing (PMI), Motivational Interviewing only (MI) or Waitlist Control (WC.) In the second, expanded phase of the study, an additional 325 peer dyads (total n = 650, ntarget client = 325, npeer = 325) will be randomized to receive either Peer-Enhanced Motivational Interviewing, Motivational Interviewing only (MI) or Waitlist Control.

DETAILED DESCRIPTION:
This project randomizes peer dyads, consisting of one Emerging Adult (EA), 18-29 years old, who both has a substance use problem and attends a Federally-qualified Health Center (i.e. target client), and one peer, to one of three conditions. In the Peer-Enhanced Motivational Interviewing (PMI) condition, target clients and peers will receive separate one-hour sessions of Motivational Interviewing (MI), an empirically-supported treatment that helps individuals work through ambivalence about making changes in substance use. MI is thought to work because it is a non-confrontational intervention where a therapist empathetically reviews substance use behaviors, listens empathetically, and reinforces any client statements indicating a desire to change. With the "peer" of each PMI dyad, the therapist presents peer with data about the extent of the target client's substance use, builds the peer's motivation to help their friend, and teaches the peer communication skills they can use to influence the target client's substance use. In the Motivational Interviewing only (MI) condition, the target client alone will receive the MI intervention with no peer participation. In the Waitlist (WC) condition, target clients and peers can receive the intervention at 2 months into the follow-up period for the PMI group.

The main purpose of this study is to test whether a Peer-Enhanced Motivational Interviewing (PMI) intervention, which has been successful with college students, results in superior alcohol and marijuana use outcomes for emerging adults (EA), ages 18-29, who are clients of Federally-qualified Health Centers, and their peers. Seventy-five peer dyads (total n = 150, ntarget client = 75, npeer = 75) will be randomized to receive either Peer-Enhanced Motivational Interviewing (PMI), Motivational Interviewing only (MI) or Waitlist Control (WC.)

ELIGIBILITY:
Inclusion Criteria:

* For the Target Client

  1. Score 5 or higher on the AUDIT-C measure and/or use alcohol or marijuana 13 days or more out of the past 90 days,
  2. Have a friend that they are willing to refer to the study to be their 'peer' (support) and that peer agrees to participate,
  3. Are able to complete baseline and follow-up assessments and have a valid email,
  4. Are willing to be video recorded, and
  5. Are fluent in English
* For the Peer

  1. Have weekly contact with the participating Target Client who referred them,
  2. Are will to attend all study procedures (i.e. baseline assessment, intervention, follow up),
  3. Are willing to be video record,
  4. Are fluent in English

Exclusion Criteria:

* For the Target Client

  1. Are current students in the lead Investigator's classes,
  2. Are seeking residential treatment at the time of the screening call,
  3. Are incarcerated or court-ordered to receive treatment at the time of the screening call,
  4. Use drugs besides marijuana or alcohol over 45 of the past 90 days.
* For the Peer

  1. Are current students in the lead Investigator's classes,
  2. Are seeking residential treatment at the time of the screening call,
  3. Are incarcerated or court-ordered to receive treatment at the time of the screening call,
  4. Use drugs besides marijuana or alcohol over 45 of the past 90 days,
  5. Are romantic partners of the Target Client

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Change: Global Appraisal of Individual Needs (GAIN) Substance Problem Scale | Baseline and at month 1, 2, 3, 6 and 9 post-intervention period
  A 16-item scale composed of lifetime symptoms of substance abuse, dependence, and substance-induced health and psychological disorders based on the Diagnostic and Statistical Manual of Mental Disorders (DSM) -IV.

SECONDARY OUTCOMES:
Change: Marijuana Consequences Questionnaire (MACQ) | Baseline and at month 1, 2, 3, 6 and 9 post-intervention period
  A 50-item self-report measure modeled after the Young Adult Alcohol Consequences Questionnaire (YAACQ) assessing marijuana problems over the past 6 months. A 6-month time frame was chosen to adequately capture potential infrequent consequences among marijuana users. Each item is rated dichotomously (yes/no) to indicate whether the marijuana-related problem occurred in the last 6 months.
Change: Days of Combined Cannabis and Alcohol Use | Baseline and at month 1, 2, 3, 6 and 9 post-intervention period
  Past month measure of days (out of past 30) when participant used both marijuana and alcohol (based on Stein et al., 2018)
Change: Days of Cannabis and Binge Alcohol Use | Baseline and at month 1, 2, 3, 6 and 9 post-intervention period
  Past month measure of days (out of past 30) of use of either substance. Binge drinking calculated from Time-Line Follow-Back (TLFB) as number of days of consuming 4+ (females)/5+ (males) drinks. Items drawn from GAIN's Substance Frequency Scale.
Change: Drinking Consequences | Baseline and at month 1, 2, 3, 6 and 9 post-intervention period
  From the Rutgers Alcohol Problems Index and used to indicate indicates the frequency of experiencing negative consequences due to alcohol use.
Change: Urine Testing | Baseline and at month 1, 2, 3, 6 and 9 post-intervention period
  National Institute of Drub Abuse-approved urine test kit to determine presence of Marijuana metabolites in urine.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas C Smith, PhD, Principal Investigator — University of Illinois Urbana Champaign School of Social Work
Locations (1):
- School of Social Work, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No